CLINICAL TRIAL: NCT00610376
Title: A Controlled Trial to Assess the Effect of a Health Promotion Intervention on Hygiene Behavior and Illness Absenteeism in Jerusalem Preschools
Brief Title: Jerusalem Handwashing Study
Acronym: JHS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hebrew University of Jerusalem (Other)
Collaborators: Ministry of Health, Israel (Other Government); Hadassah Medical Organization (Other); Israel National Institute for Health Policy and Health Services Research (Other Government); Ministry of Education, Israel (Other Government); Municipality of Jerusalem, Israel (Unknown)
Responsible Party: Laura (Leah) Rosen, Hebrew University, Israel (at the time of conduct of the trial)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JHS1; NIHP Doctoral Stipend [m-2-02]
Record Dates: First submitted 2008-01-27; First posted 2008-02-08 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2008-01

CONDITIONS: Illness Absenteeism; Handwashing Behavior
Keywords: Handwashing; Randomized controlled trial; Cluster randomization; Community intervention trial; Disease prevention; Pediatric communicable disease; Preschool; Illness absenteeism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1A (Experimental): Preschools randomized to this group received a multicomponent intervention to improve handwashing behavior of the children. Children within the preschool intervention group were individually randomized to a home intervention or a home control intervention program. The children in this arm received the home intervention component.
  Interventions: Behavioral: Preschool handwashing intervention program; Behavioral: Home component intervention
- 2 (Active Comparator): This group did not receive any special treatment during the study, but did receive the intervention at the close of the study
  Interventions: Behavioral: Preschool handwashing intervention program
- 1B (Experimental): Preschools randomized to this group received a multicomponent intervention to improve handwashing behavior of the children. Children within the preschool intervention group were individually randomized to a home intervention or a home control intervention program. The children in this arm received the home control component.
  Interventions: Behavioral: Preschool handwashing intervention program; Behavioral: Home component intervention

INTERVENTIONS:
Behavioral: Preschool handwashing intervention program — This preschool-based intervention program used a multi-pronged approach that included elements aimed at preschool staff, children, and school nurses, as well as hygienic changes to the classroom environment.
Behavioral: Home component intervention — The home component was intended to reinforce handwashing practices through education in the home. It consisted of a video, a magnet, and a card.
  Arms: 1A; 1B

SUMMARY:
The primary objective of this preschool intervention trial was to determine whether a hygiene program can promote handwashing and thereby reduce illness absenteeism.

DETAILED DESCRIPTION:
Please see citations of published reports.

ELIGIBILITY:
Inclusion Criteria:

* Preschool teachers of 3- and 4-year-old children in the state-run public system of the Jerusalem region, who were recommended by their supervisors as being likely to comply with the protocol.

Exclusion Criteria:

* Exposure to project during testing phase (N=1 preschool), preschool which included new Ethiopian immigrants who were unlikely to have phones or speak Hebrew (N=1 preschool)
* Project staff knew teachers personally and thought they would not comply with protocol (N=2 teachers).

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1029 (Actual)
Dates: Start 2000-09; Primary Completion 2001-12 (Actual); Study Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Illness absenteeism | Each school day during study period

SECONDARY OUTCOMES:
Handwashing behavior | Observational visits in classrooms (3-4)

CONTACTS AND LOCATIONS:
Overall Officials: Laura J Rosen, PhD, Principal Investigator — Hebrew University (at time of study); David M Zucker, PhD, Principal Investigator — Hebrew University; Orly Manor, PhD, Principal Investigator — Hebrew University; Dan Engelhard, MD, Principal Investigator — Hadassah Hebrew Univeristy Hospital
Locations (1):
- Hebrew University, Jerusalem, Israel

REFERENCES:
- [Background] Rosen L, Manor O, Engelhard D, Brody D, Rosen B, Peleg H, Meir M, Zucker D. Can a handwashing intervention make a difference? Results from a randomized controlled trial in Jerusalem preschools. Prev Med. 2006 Jan;42(1):27-32. doi: 10.1016/j.ypmed.2005.09.012. Epub 2005 Nov 21. PMID 16300823
- [Background] Rosen L, Manor O, Engelhard D, Zucker D. Design of the Jerusalem Handwashing Study: meeting the challenges of a preschool-based public health intervention trial. Clin Trials. 2006;3(4):376-84. doi: 10.1177/1740774506070690. PMID 17060212
- [Background] Rosen L, Manor O, Engelhard D, Zucker D. In defense of the randomized controlled trial for health promotion research. Am J Public Health. 2006 Jul;96(7):1181-6. doi: 10.2105/AJPH.2004.061713. Epub 2006 May 30. PMID 16735622